CLINICAL TRIAL: NCT06743126
Title: A Prospective, Multicenter, Open-label, Randomized, Actively Controlled, Parallel-group Phase 3 Clinical Trial to Evaluate Efficacy, Safety, and Tolerability of IMA203 Versus Investigator's Choice of Treatment in Patients With Previously Treated, Unresectable or Metastatic Cutaneous Melanoma (ACTengine® IMA203-301)
Brief Title: SUPRAME-ACTengine® IMA203 vs. Investigator's Choice of Treatment in Previously Treated, Unresectable or Metastatic Cutaneous Melanoma
Acronym: SUPRAME
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Immatics US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMA203-301
Record Dates: First submitted 2024-12-11; First posted 2024-12-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Melanoma, Cutaneous Malignant
MeSH Terms: conditions — Melanoma, Cutaneous Malignant | interventions — Nivolumab; relatlimab; Opdualag; lifileucel; pembrolizumab; Ipilimumab; Dacarbazine; Temozolomide; Paclitaxel; Carboplatin; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Non-myeloablative chemotherapy for lymphodepletion (LD) over 4 days using fludarabine (FLU) and cyclophosphamide (CY), one-time administration of IMA203, and adjunctive therapy with low dose interleukin (IL)-2 for up to 10 days, starting approximately 24 h after IMA203 infusion, optional bridging therapy
  Interventions: Biological: IMA203
- Control arm- investigator's choice (Active Comparator): Investigator's choice of treatment approved by the respective Competent Authority (nivolumab plus relatlimab [Opdualag®], lifileucel, nivolumab, pembrolizumab, ipilimumab, or chemotherapy [e.g., dacarbazine, temozolomide, paclitaxel, alb-bound paclitaxel, or paclitaxel plus carboplatin]) as determined by the site investigator in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC), optional bridging therapy.
  Interventions: Biological: nivolumab plus relatlimab; Biological: lifileucel; Biological: nivolumab; Biological: pembrolizumab; Biological: ipilimumab; Drug: Dacarbazine; Drug: temozolomide; Drug: paclitaxel; Drug: paclitaxel plus carboplatin; Drug: Albumin-Bound Paclitaxel

INTERVENTIONS:
Biological: IMA203 — one-time administration of IMA203, and adjunctive therapy with low dose interleukin (IL)-2 for up to 10 days, starting approximately 24 h after IMA203 infusion, optional bridging therapy
  Other Names: anzutresgene autoleucel; anzu-cel
  Arms: Experimental arm
Biological: nivolumab plus relatlimab — in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC)
  Other Names: Opdualag®
  Arms: Control arm- investigator's choice
Biological: lifileucel — in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC)
  Other Names: AMTAGVI
  Arms: Control arm- investigator's choice
Biological: nivolumab — in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC)
  Other Names: Opdivo®
  Arms: Control arm- investigator's choice
Biological: pembrolizumab — in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC)
  Other Names: Keytruda®
  Arms: Control arm- investigator's choice
Biological: ipilimumab — in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC)
  Other Names: Yervoy
  Arms: Control arm- investigator's choice
Drug: Dacarbazine — in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC)
  Other Names: DTIC-Dome
  Arms: Control arm- investigator's choice
Drug: temozolomide — in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC)
  Other Names: Temodar
  Arms: Control arm- investigator's choice
Drug: paclitaxel — in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC)
  Other Names: Taxol
  Arms: Control arm- investigator's choice
Drug: paclitaxel plus carboplatin — in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC)
  Other Names: Carbo/Taxol®
  Arms: Control arm- investigator's choice
Drug: Albumin-Bound Paclitaxel — in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC)
  Other Names: Abraxane®
  Arms: Control arm- investigator's choice

SUMMARY:
This clinical trial is a prospective, multicenter, open-label, randomized, actively controlled, parallel-group Phase 3 clinical trial to evaluate the efficacy, safety and tolerability of treatment with IMA203 administered at the recommended phase 2 dose versus investigator's choice of treatment in patients with previously treated, unresectable or metastatic cutaneous melanoma.

DETAILED DESCRIPTION:
SCREENING: Patient eligibility will be determined by protocol inclusion/exclusion criteria including HLA (human leukocyte antigen) screening. Leukapheresis for potential manufacturing of the IMA203 cellular product may be performed, if patients are HLA-A*02:01 positive and meet the eligibility criteria for leukapheresis.

MANUFACTURING: IMA203 products will be made from the patients' white blood cells.

TREATMENT- Experimental arm: Lymphodepletion with cyclophosphamide and fludarabine will occur in the days before the IMA203 product infusion to improve the duration of time that IMA203 product stays in the body. The patient will be admitted to the hospital during the T-cell infusion.

After the IMA203 product infusion, a low dose of IL-2 will be given subcutaneously for up to 10 days.

TREATMENT- Control arm: Investigator's choice of treatment approved by the respective competent authority (nivolumab plus relatlimab [Opdualag®], lifileucel, nivolumab, pembrolizumab, ipilimumab, or chemotherapy [e.g., dacarbazine, temozolomide, paclitaxel, alb-bound paclitaxel, or paclitaxel plus carboplatin]) as determined by the site investigator in accordance with current respective prescribing information (PI) and/or summary of product characteristics (SmPC).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed and documented cutaneous melanoma- CM patients (including acral melanoma) with unresectable or metastatic disease
* HLA-A*02:01 positive
* Adequate selected organ function per protocol
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Disease progression (resistance, toxicity) on or after at least one PD-1 inhibitor, applied either as monotherapy or in combination with other therapies as treatment for unresectable or metastatic cutaneous melanoma
* Patients with BRAF mutation should have been treated with one prior line of BRAF-directed therapy (with or without a MEK inhibitor) prior to initial eligibility assessment, unless deemed not clinically indicated at Investigator's discretion due to concurrent medical condition, prior toxicity, or if declined by the patient
* Life expectancy more than 6 months
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
* Female patient of childbearing potential must use adequate contraception from randomization until 12 months after the infusion of IMA203 or in line with the instructions provided for investigator's choice treatment (in the control arm)
* Male patient must agree to use effective contraception or be abstinent while on study and for 6 months after the infusion of IMA203 or in line with the instructions provided for investigator's choice treatment (in the control arm)
* The patient must have recovered from any side effects of prior therapy to Grade 1 or lower prior to randomization.

Exclusion Criteria:

* Primary mucosal or uveal melanoma and melanoma of unknown primary
* History of other malignancies (except for adequately treated basal or squamous cell carcinoma or carcinoma in situ) within the last 3 years
* Serious autoimmune disease Note: At the discretion of the investigator, these patients may be included if their disease is well controlled without the use of immunosuppressive agents.
* History of cardiac conditions as per protocol
* Prior allogenic stem cell transplantation or solid organ transplantation
* Concurrent severe and/or uncontrolled medical disease that could compromise participation in the study
* History of or current immunodeficiency disease or prior treatment compromising immune function at the discretion of the treating physician
* History of hypersensitivity to CY, FLU, or IL-2 or presence of any contraindications and other limitations for planned treatment with investigator's choice as laid down in the current versions of the respective PIs / SmPCs
* Known hypersensitivity to any of the rescue medications
* History of or current immunodeficiency disease or prior treatment compromising immune function at the discretion of the investigator
* Positive for HIV infection or with active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection.
* Any condition contraindicating leukapheresis
* Pregnant or breastfeeding
* Any other condition that would, in the investigator's or sponsor's judgment, contraindicate the patient's participation in the clinical trial because of safety concerns or compliance with clinical trial procedures (e.g., psychiatric disorders or substance dependence, neurological impairment)
* Patient has received systemic corticosteroids within 2 weeks prior to leukapheresis,
* Patient has received surgery or other anti-cancer therapies, any agent that is likely to suppress bone marrow function, or investigational medicinal products within 7 days prior to leukapheresis.
* Patients with any active infection or ongoing reactivation of infection
* Patients who underwent non-myeloablative lymphodepletion prior to cell therapy within the last 6 months
* Prior treatment with IMA203
* Patients with ascites, pleural or pericardial effusion which requires repeated (2 within 4 weeks) or continuous paracentesis, thoracentesis or pericardiocentesis within last 2 months
* Patients with LDH greater than 2.0-fold ULN
* Concurrent treatment in another clinical trial or a device study that could interfere with the IMA203 treatment or planned investigator's choice treatment
* Patients with active brain metastases or leptomeningeal metastases
* Patient has received any investigational therapies, inactivated vaccines, chronic use of systemic corticosteroids or IV antibiotics within 1 week prior to randomization, or live vaccines within 4 weeks prior to randomization
* Patient has received any anti-cancer therapy (prior anti-cancer treatment or bridging therapy) or radiotherapy within 1 week prior to start of trial treatment
* Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival assessed by BICR | up to 5 years post first treatment of last patient
  progression-free survival (PFS), centrally assessed (by blinded independent central review) using RECIST 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years post first treatment of last patient
  conducted onsite or can be performed by phone
Objective response rate (ORR) | up to 5 years post first treatment of last patient
  complete responses (CR) and partial response (PR) based on best overall response (BOR), locally and centrally (by blinded independent central review) assessed using RECIST 1.1
Progression-free survival | up to 5 years post first treatment of last patient
  Progression-free survival locally assessed using RECIST 1.1
Treatment-emergent adverse events (TEAEs) | until 85 days after cell therapy treatment or 30 days after last treatment
  To evaluate safety and tolerability of treatment with IMA203 compared with control (investigator's choice)
Adverse events of special interest (AESIs) | until 85 days after cell therapy treatment or 30 days after last treatment
  To evaluate safety and tolerability of treatment with IMA203 compared with control (investigator's choice)
Treatment-emergent serious adverse events (TESAEs) | until 85 days after cell therapy treatment or 30 days after last treatment
  To evaluate safety and tolerability of treatment with IMA203 compared with control (investigator's choice)
Frequency and duration of dose interruptions, reductions, and discontinuations | up to 5 years post first treatment of last patient
  To evaluate safety and tolerability of treatment with IMA203 compared with control (investigator's choice)
EORTC QLQ-C30 | up to 5 years post first treatment of last patient
  To evaluate the patient-reported quality of life before and after treatment with IMA203 compared with control (investigator's choice)
EQ-5D-5L | up to 5 years post first treatment of last patient
  To evaluate the patient-reported quality of life before and after treatment with IMA203 compared with control (investigator's choice)

CONTACTS AND LOCATIONS:
Overall Officials: Cedrik Britten, M.D., Study Director — Immatics US, Inc.
Locations (51):
- United States (38):
  - Mayo Clinic, Phoenix, Arizona
  - Honor Health Research Institute, Scottsdale, Arizona
  - City of Hope National Medical Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - The University of Colorado, Anschutz Medical Campus, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami - Sylvester Comprehensive Cancer Cente, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - University of MD Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Atlantic Health System/Morristown Medical Center, Morristown, New Jersey
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - UNC Hospitals, The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Taussig Cancer Institute, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jeffersion University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - SCRI Oncology Partners, Nashville, Tennessee
  - Baylor University, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Germany (12):
  - Universitatsklinikum Koeln, Cologne, Northrhine-W Estphalia
  - Charite Universitaetsmedizin Berlin KöR, Berlin
  - Universitaetsklinikum Bonn AöR, Bonn
  - University Hospital Cologne AöR, Cologne
  - Technische Universitaet Dresden, Dresden
  - Universitaetsklinikum Erlangen AöR, Erlangen
  - Universitaetsklinikum Essen AöR, Essen
  - Goethe University Frankfurt, Frankfurt am Main
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Universitaetsklinikum Heidelberg AöR, Heidelberg
  - Universitaet Leipzig, Leipzig
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KöR, Mainz